CLINICAL TRIAL: NCT00806572
Title: Phase II Multiple Dose Treatment of Type 1 Diabetes Mellitus With hOKT3gamma1(Ala-Ala)
Brief Title: Treatment With hOKT3gamma1(Ala-Ala) in T1DM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Adverse events related to drug lot
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN007AI; NDB01
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes, juvenile diabetes, teplizumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — teplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: hOKT3gamma1(Ala-Ala)
- Control (No Intervention)

INTERVENTIONS:
Drug: hOKT3gamma1(Ala-Ala) — 3 cycles, six months apart, each consisting of 12 daily infusions with 455-1818ug/m2 hOKT3g1(Ala-Ala)
  Other Names: teplizumab
  Arms: Treatment

SUMMARY:
This is a phase II study to examine the clinical and immunological effects of humanized FcR non-binding anti-CD3 mAb in participants with Type 1 diabetes mellitus (T1DM), and to develop this therapy to prevent the immune destruction leading to β cell loss.

DETAILED DESCRIPTION:
This is a 2-arm, open-label phase II trial involving 0 or 3 cycles of treatment 6 months apart with hOKT3γ1 (Ala-Ala), over the first year of disease in participants with new onset T1DM. Each cycle consists of 12 daily doses of hOKT3γ1 (Ala-Ala).

Participants will be randomized in a ratio of 2:1 to either the experimental arm or the control arm and will be stratified by study site.

To be eligible, participants must be: male or female between 7-30 years of age, diagnosed with T1DM within the past 6 weeks, have a body weight ≥26 kg at the time of enrollment and have detectable anti-GAD, anti-ICA512/IA-2, or insulin autoantibodies (if the participant has been on insulin ≤10 days).

Participants randomized to the experimental group will start the first cycle of hOKT3γ1 (Ala-Ala) within 4-8 weeks of T1DM diagnosis. Each participant randomized to the experimental group will receive 3 cycles of drug treatment, separated by 6 months each. Each cycle consists of 12 days of drug treatment.

Both groups will undergo the Mixed Meal Stimulated C-Peptide Test and receive blood draws for mechanistic studies on the same schedule.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with T1DM within the past 6 weeks
* have a body weight ≥26 kg at the time of enrollment
* have detectable anti-GAD, anti-ICA512/IA-2, or insulin autoantibodies (if the participant has been on insulin ≤10 days).

Exclusion Criteria:

* Pregnant or lactating females;
* Prior OKT3 treatment;
* Known hypersensitivity to murine products;
* Uncompensated heart failure or fluid overload, recent myocardial infarction;
* History of epilepsy, cancer, active infection, atopic disease, active Grave's disease, cystic fibrosis, sickle cell anemia, neuropathy, peripheral vascular disease, cerebrovascular disease, any concurrent autoimmune diseases, asthma;
* Any medical condition that in the opinion of the investigator will interfere with safe completion of the trial;
* Inability to give informed consent;
* Prior participation in a clinical trial that could potentially affect diabetes or immunologic status;
* Participation in a clinical trial within the last 6 weeks;
* HIV positive;
* Positive for Hepatitis B surface antigen or Anti-Hepatitis C antibody;
* Seropositivity for Toxoplasmosis (IgG);
* Lymphopenia (<1000 lymphocytes/microliter);
* Thrombocytopenia (<150,000/mm3 platelets);
* Anemia (Hgb < 10g/dL);
* Vaccination with a live virus within the past 6 weeks;
* Positive PPD skin test;
* Any infectious mononucleosis-like illness within the 3 months prior to enrollment;
* Serologic evidence of acute infection with EBV or CMV based on tests listed and as defined by the protocol.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2002-05; Primary Completion 2004-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
4-hour C-peptide AUC | 24 months

SECONDARY OUTCOMES:
Insulin usage | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kevan C Herold, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Naomie Berrie Diabetes Center, Columbia University, New York, New York
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in Participant level data and additional relevant materials are available to the public in : 1.) the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers; and 2.) TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal that makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Result] Herold KC, Gitelman S, Greenbaum C, Puck J, Hagopian W, Gottlieb P, Sayre P, Bianchine P, Wong E, Seyfert-Margolis V, Bourcier K, Bluestone JA; Immune Tolerance Network ITN007AI Study Group. Treatment of patients with new onset Type 1 diabetes with a single course of anti-CD3 mAb Teplizumab preserves insulin production for up to 5 years. Clin Immunol. 2009 Aug;132(2):166-73. doi: 10.1016/j.clim.2009.04.007. Epub 2009 May 14. PMID 19443276
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: ITN007AI-NDB01 — http://www.itntrialshare.org/project/Studies/ITN007AIPUBLIC/Study%20Data/begin.view? — TrialShare is a portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.Creating an account for ITN TrialShare is free and allows for searching studies of interest.
- Available data/document: Study protocol synopsis, -navigator, -schedule of events,-data &reports, -specimens et al.: ITN007AI-NDB01 — http://www.itntrialshare.org/project/Studies/ITN007AIPUBLIC/Study%20Data/begin.view? — TrialShare is a portal developed by the Immune Tolerance Network (ITN) that makes data from the consortium's clinical trials publicly available without charge.Creating an account for ITN TrialShare is free and allows for searching studies of interest.
- Available data/document: Individual Participant Data Set: SDY569 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY569 — ImmPort study identifier is SDY569. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.
- Available data/document: Study summary, -design, -medications, -demographics, -lab tests, and -files.: SDY569 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY569 — ImmPort study identifier is SDY569. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts and is available to the Public.